CLINICAL TRIAL: NCT05731817
Title: Profile of COVID-19 Patients Related to Fatigue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Torres Sánchez, PT, PhD, Principal investigator, Universidad de Granada
Other Study IDs: COVIDATE-01
Record Dates: First submitted 2023-02-10; First posted 2023-02-16 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: COVID-19; fatigue
MeSH Terms: conditions — COVID-19; Fatigue | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: COVID-19 patients
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — N/A - observational study.

SUMMARY:
More than half of recovered COVID-19 patients experience fatigue. Studies are needed to define the profile of these patients.

The objective of this study is to evaluate the profile of surviving patients of COVID-19 in relation to fatigue.

DETAILED DESCRIPTION:
Background: More than half of recovered COVID-19 patients experience fatigue. Studies are needed to define the profile of these patients.

Objectives: Evaluate the profile of surviving patients of COVID-19 in relation to fatigue;

Methodology: Observational study. The profile of the survivors of COVID-19 will be described, dividing them into 2 groups based on the presence or absence of fatigue.

Patients will be recruited from the Virgen de las Nieves University Hospital in Granada.

The evaluation will be carried out through Google forms, telematic means or face-to-face depending on the variables.

A symptomatic evaluation of fatigue, aspects related to fatigue and physical performance will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COVID-19
* adults (>18 years)
* basic knowledge and access to the internet
* wish to participate in the study and sign the informed consent

Exclusion Criteria:

* patients with severe comorbidities that interfere with the ability to perform the study, and those with mental, physical or organic problems that under medical criteria may pose a risk to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients
Sampling Method: Non-Probability Sample
Enrollment: 398 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Fatigue | Through study completion, an average of 1 year
  To assess perceived fatigue using the borg modified scale. Scale ranges from 0 to 10, with higher punctuation indicating higher fatigue perception.
Multidimensional Fatigue | Through study completion, an average of 1 year
  To assess multidimensional fatigue using the multidimensional fatigue inventory
Fatigue Severity | Through study completion, an average of 1 year
  To assess fatigue severity using the fatigue severity scale. The total score ranges from 7 to 63 points, with higher punctuation indicating higher fatigue severity
Fatigue Impact | Through study completion, an average of 1 year
  To assess fatigue impact using the modified fatigue impact scale. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities. This scale can range from 0 to 36.
Muscular Fatigue | Through study completion, an average of 1 year
  To assess muscular fatigue using surface electromyography

SECONDARY OUTCOMES:
COVID-19 information | Through study completion, an average of 1 year
  To assess information about the date and symptoms when COVID-19 was diagnosed
Dyspnea | Through study completion, an average of 1 year
  To assess Dyspnea perception using the borg modified scale
Cough | Through study completion, an average of 1 year
  To assess cough using the leicester cough questionnaire
Pain intensity | Through study completion, an average of 1 year
  To assess pain intensity using the visual analogue scale and brief pain inventory
Functional status | Through study completion, an average of 1 year
  To assess functional status using the post-covid functional scale and functional independence measure
Frailty | Through study completion, an average of 1 year
  To assess frailty using the clinical frailty scale
Health-related Quality of life | Through study completion, an average of 1 year
  To assess health-related quality of life using the euroqol-5d
Psychological status | Through study completion, an average of 1 year
  To assess Psychological status using the hospital anxiety and depression scale
Sleep quality | Through study completion, an average of 1 year
  To assess sleep quality using the Pittsburgh Sleep Quality Index
Nutritional status | Through study completion, an average of 1 year
  To assess nutritional status using the mini nutritional assessment
Physical activity | Through study completion, an average of 1 year
  To assess physical activity using the international physical activity questionnaire. This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in Metabolic Equivalent (MET)-min/week and time spent sitting.
Kinesiophobia | Through study completion, an average of 1 year
  To assess kinesiophobia using the TAMPA scale
Exercise capacity | Through study completion, an average of 1 year
  To assess exercise capacity using the Short Physical Performance Battery and the 6 minutes walk test
Strength | Through study completion, an average of 1 year
  To assess strength using dynamometry
Heart rate variability | Through study completion, an average of 1 year
  To assess heart rate variability using holter

CONTACTS AND LOCATIONS:
Overall Officials: Irene Torres Sánchez, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Spain

REFERENCES:
- [Derived] Perez-Gisbert L, Morales-Garcia C, Sanchez-Martinez JA, Gonzalez-Gutierrez MV, Valenza MC, Torres-Sanchez I. Severity Matters: How COVID-19 Severity Impacts Long-Term Effects on Symptoms, Physical Activity and Functionality-An Observational Study. Healthcare (Basel). 2025 Feb 6;13(3):333. doi: 10.3390/healthcare13030333. PMID 39942522